CLINICAL TRIAL: NCT01431157
Title: Effects of Nocturnal Nasal Oxygen on Biomarkers in Sleep Apnea Patients With Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen Gottlieb, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP-00049080
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Sleep Apnea; Heart Failure
Keywords: Sleep Apnea Syndrome; Heart Failure; Oxygen Inhalation Therapy
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal oxygen (Active Comparator): Nocturnal nasal oxygen
  Interventions: Procedure: Nocturnal nasal oxygen
- No nasal oxygen (Placebo Comparator)
  Interventions: Other: No nasal oxygen

INTERVENTIONS:
Procedure: Nocturnal nasal oxygen — Nasal oxygen at 2 l/min will be given at night
  Arms: Nasal oxygen
Other: No nasal oxygen — Patients will have no intervention for sleep apnea
  Arms: No nasal oxygen

SUMMARY:
Sleep apnea syndrome is clinically defined by frequent pauses in breathing during sleep and symptoms, such as being tired. It can decrease the restfulness of sleep and decreases the level of oxygen in the blood. Sleep apnea patients suffer from daytime sleepiness, hypertension, coronary artery disease (CAD), stroke, ischemic heart disease, arrhythmias, pulmonary hypertension, heart failure, and premature death. There is significant evidence suggesting that nighttime decreases in blood oxygen levels are the primary cause of many of the abnormalities associated with this disease.

Epidemiological studies have demonstrated a surprisingly high prevalence of sleep apnea. Mild sleep apnea is present in 17% of adults in the general population and moderate to severe sleep apnea is present in 5.7% of adults. Among patients with heart failure the prevalence skyrockets. Multiple studies have found the prevalence of moderate to severe sleep apnea to be anywhere from 11-53% in heart failure patients.

Continuous positive airway pressure (CPAP) therapy is currently the standard of care for sleep apnea sufferers regardless of the severity of their disease. In patients without heart failure, CPAP therapy has numerous benefits and several long term studies have reported that CPAP causes less cardiovascular disease as well as a long term improvement in cardiovascular symptoms and mortality among patient with severe sleep apnea.

In heart failure patients, CPAP has shown some beneficial short term effects but evidence of long term improvements in symptoms and mortality are lacking. Compliance with CPAP therapy reduces systolic blood pressure, improves cardiac function, raises oxygen levels, and increases exercise tolerance. On the other hand, CPAP has not been shown to affect survival or number of hospitalizations in heart failure patients. Moreover, compliance with CPAP is often poor and many people cannot tolerate it. This further limits the therapeutic effectiveness of this intervention.

The purpose of this study is to assess whether nocturnal oxygen administration via nasal cannula alone can improve outcomes in congestive heart failure patients with moderate to severe sleep apnea. The effects of nocturnal oxygen administration will be assessed by using biomarkers of heart stress and markers of whole body inflammation.

ELIGIBILITY:
Inclusion Criteria:

* RDI > 15
* Symptomatic Heart failure
* Oxygen saturation < 88% during apnea
* Not currently be on nocturnal oxygen therapy, CPAP, or other PAP therapy

Exclusion Criteria:

* Hypoxemia requiring oxygen supplementation
* serum creatinine > 2.5 or on chronic dialysis
* blood pressure > 160
* pregnant
* chronic physical disability that would prevent subjects from participating in any aspect of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
BNP (a blood test which is a biomarker for heart failure) | 1 month

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baltimore VA Medical Center, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland